CLINICAL TRIAL: NCT00521846
Title: ExploR™ Modular Radial Head Data Collection
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Donald Lee, Professor of Orthopaedic Surgery, Vanderbilt University Medical Center
Other Study IDs: 070155
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Elbow Fracture
MeSH Terms: conditions — Elbow Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- 1: As part of their routine care, patient's will receive Biomet modular radial head replacement. This study is an observational, prospective study that monitors the patient's pain, functional ability, and patient-reported outcomes.
  Interventions: Device: Biomet Explor Modular Radial Head Replacement

INTERVENTIONS:
Device: Biomet Explor Modular Radial Head Replacement — As part of the patient's routine care, they will undergo a radial head replacement using the Biomet Explor Modular Radial Head system.

SUMMARY:
The purpose of this prospective clinical data collection is to document the performance and clinical outcomes of the ExploR Modular Radial Head.

DETAILED DESCRIPTION:
The purpose of this prospective clinical data collection is to document the performance and clinical outcomes of the ExploR Modular Radial Head.

The radial head on which data will be collected is legally marketed and is not investigational or experimental. This data collection effort will document the clinical outcomes of the radial head.

Surgical techniques and patient care are to be standard for the surgeon participating in the protocol. There will be no experimental or investigational surgical techniques used. The devices and products are to be used in accordance with their instructions for use and/or approved labeling.

The outcomes and data collected include:

The Mayo Clinic Performance Index for The Elbow The Quick DASH Outcome Measure Radiographic Evaluation

All revisions, complications, and adverse events will also be recorded. Inclusion Criteria

Replacement of the radial head for degenerative or post-traumatic disabilities presenting pain, crepitation, and decreased motion at the radio-humeral and/or proximal radio-ulnar joint with:

1. Joint destruction and/or subluxation visible on x-ray
2. Resistance to conservative treatment Primary replacement after fracture of the radial head Symptomatic sequelae after radial head resection Revision following failed radial head arthroplasty

Patient selection factors to be considered:

1. Need to obtain pain relief and improve function
2. Ability and willingness of the patient to follow instructions, including control of weight and activity levels
3. A good nutritional state of the patient
4. The patient must have reached full skeletal maturity

Exclusion Criteria Patients who have infection, sepsis, and osteomyelitis Patients who are uncooperative or have neurologic disorders who is capable or unwilling to follow directions Patients with distant foci of infections which may spread to the implant site Patients with rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram Patients who are pregnant Patients who are under 18 years of age Patients who have had fractures of the humerus Patients who have had revisions where other devices and treatments have failed

ELIGIBILITY:
Inclusion Criteria

Replacement of the radial head for degenerative or post-traumatic disabilities presenting pain, crepitation, and decreased motion at the radio-humeral and/or proximal radio-ulnar joint with:

1. Joint destruction and/or subluxation visible on x-ray
2. Resistance to conservative treatment Primary replacement after fracture of the radial head Symptomatic sequelae after radial head resection Revision following failed radial head arthroplasty

Patient selection factors to be considered:

1. Need to obtain pain relief and improve function
2. Ability and willingness of the patient to follow instructions, including control of weight and activity levels
3. A good nutritional state of the patient
4. The patient must have reached full skeletal maturity

Exclusion Criteria Patients who have infection, sepsis, and osteomyelitis Patients who are uncooperative or have neurologic disorders who is capable or unwilling to follow directions Patients with distant foci of infections which may spread to the implant site Patients with rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram Patients who are pregnant Patients who are under 18 years of age Patients who have had fractures of the humerus Patients who have had revisions where other devices and treatments have failed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be any individual that seeks care at Vanderbilt University Medical Center for a radial head fracture/dislocation that requires replacement using a Biomet Explor Modular Radial Head implant (routine care).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
We will measure the performance and clinical outcomes of the ExploR Modular Radial Head based on data collection from the following forms: The Mayo Clinic Performance Index for The Elbow, The Quick DASH Outcome Measure, Radiographic Evaluation | 5 years
Patient examination measurements and radiographic measurements will be used to determine the effects of the Modular Radial Head implant. | Pre-op, 6 week, 3 months, 6 months, 1 year, 2 year, 3 year, 4 year, 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Donald H Lee, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Will not be shared.